CLINICAL TRIAL: NCT01330524
Title: Comparison of Intravitreal Bevacizumab and Triamcinolone With Placebo in Acute Nonarteritic Anterior Ischemic Optic Neuropathy
Brief Title: Comparison of Intravitreal Bevacizumab and Triamcinolone With Placebo
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: morteza entezari, Ophthalmic Research center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8749
Record Dates: First submitted 2011-03-08; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2009-11

CONDITIONS: Acute Nonarteritic Anterior Ischemic Optic Neuropathy
MeSH Terms: interventions — Bevacizumab; Triamcinolone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Avastin and Triamcinolone (Active Comparator)
  Interventions: Drug: Avastin and Triamcinolone
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Avastin and Triamcinolone — 1.25 mg Avastin and 2mg Triamcinolone will be injected trough vitreal
  Arms: Avastin and Triamcinolone
Other: placebo — 2mg placebo
  Arms: Placebo

SUMMARY:
In this study 16 Patients diagnosed with Nonarteritic Anterior Ischemic Optic Neuropathy(NSION) who had a sudden mono ocular vision loss associated with optic disc edema and positive Marcus Gunn in less than 30 days without exclusion criteria are randomly divided in two groups 1) control 2) case. In case group Avastin and Triamcinolone will be injected trough vitreal and placebo will be injected in control group. BCVA and Visual field will be then measured in these two groups.

ELIGIBILITY:
Inclusion criteria:

* Sudden mono ocular vision loss associated with optic disc edema and positive Marcus Gunn (<30 days)

Exclusion criteria:

* Any eye disease except NAION(Nonarteritic Anterior Ischemic Optic Neuropathy)
* Neurologic defect
* Abnormal ESR, CRP, any history of retina or vitreal surgery
* Severe corneal opacity which makes retina examination impossible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Changes of Best corrected visual acuity(BCVA) | 6 month
  outcome method of measurement: Snellen chart

SECONDARY OUTCOMES:
Changes of Visual Field | 6 month
  Automated perimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Iran